CLINICAL TRIAL: NCT00932269
Title: Seroimmunity 2007. Serological Study of the Swedish Population Regarding Vaccine Preventable Diseases Within the National Immunization Program (NIP), and a Sub Study Focusing on Foreign Born 14-16 Year-Olds.
Brief Title: Seroimmunity 2007 and Sub Study of the Swedish Population Regarding Vaccine Preventable Disease
Acronym: Sero 2007
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Swedish Institute for Infectious Disease Control (Other)
Responsible Party: Assoc. Prof. Rigmor Thorstensson, Swedish Institute for Infectious Disease Control
Other Study IDs: 2007/132-31/4//2008/164-32
Record Dates: First submitted 2009-06-30; First posted 2009-07-03 (Estimated); Last update posted 2009-07-03 (Estimated); Status verified 2009-07

CONDITIONS: Diphtheria; Tetanus; Pertussis; Polio; Haemophilus Influenzae Type B; Measles; Mumps; Rubella; Hepatitis B
Keywords: Diphtheria; Tetanus; Pertussis; Polio; Haemophilus influenzae type B; Hib; Measles; Mumps; Rubella; Hepatitis B; Vaccine; Vaccination; Immunity; Vaccination program; Sweden; ELISA
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Poliomyelitis; Haemophilus Infections; Measles; Mumps; Rubella; Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Seroimmunity 2007: Cord blood from 400 newborns, 1800 children (2 - 18 years) and 2400 adults (above 18 years), randomly selected and stratified in age groups, from which blood samples are taken.
- Sub Study: 800 immigrated children (14 - 16 years) from which blood samples are taken.

SUMMARY:
This is a randomized cross-sectional study of the Swedish population. Blood samples will be collected from a subpopulation in order to estimate the age specific sero-prevalence of the Swedish population for diseases included in the National Immunization Program (NIP), and to affirm the population's protection against polio. To be able to recommend complementary immunizations to immigrated children, a sub study focusing on foreign born teenagers will also be done and compared to children of the same age born in Sweden.

DETAILED DESCRIPTION:
Besides the main objectives stated in the summary, the study consists of:

Vaccine related objectives:

* To estimate the seroprevalence regarding vaccine preventable diseases in the cohort of children about to enter adulthood (as a "receipt" of the vaccination program's functionality), and thereby form a basis for decision-making regarding recommendations about continuous vaccination in adult age
* To evaluate the concentration of antibodies that full-term newborns receive from their mothers, and to estimate plausible consequences to optimize the schedule of the NIP for each vaccine preventable disease
* To, in different age groups, evaluate changes over time and concentration of antibodies compared to a study conducted in 1997
* To evaluate plausible changes in the seroprevalence, for instance among children, related to an increased use of combined vaccines
* To document the age-specific seroprevalence against other diseases that will be vaccine preventable before start-up of new vaccination program
* To estimate the population seroprevalence against certain diseases against which vaccines have been developed during recent years and that might be introduced into the vaccination program within a couple of decades

Method:

* Adults: one blood sample of 10 mL blood from vein in arm from each individual
* Children: one blood sample of 5-10 mL blood from vein or capillary in arm from each individual
* Cord blood: one blood sample of 10 mL cord blood will be collected from each newborn in connection with childbirth

The objectives of the sub study are:

* To conduct the same type of analysis on foreign born 14-16 year olds as on 14-16 year olds being born in Sweden
* To also examine the immunity and infection situation with regard to Hepatitis B
* To conduct the corresponding examinations and priorities among the 14-16 year olds born in Sweden serving as control group

ELIGIBILITY:
Inclusion Criteria:

* informed written consent (both groups)
* immigrated to Sweden after 6 years of age from a country with polio vaccination coverage < 85 % (Sub study group)
* living and attending school in Stockholm, Gothenburg or Malmoe (Sub study group)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Seroimmunity 2007: the Swedish population.
  Sub study: foreign born children between 14-16 years of age.
Sampling Method: Probability Sample
Enrollment: 5400 (Estimated)
Dates: Start 2007-03; Primary Completion 2008-05 (Actual); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Establishing the immunity situation among specific population groups, concerning diseases targeted by the NIP, by measuring antibody levels in serum using methods In-house ELISAs, Neutralization test (NT) and ELISAs from Dade Behring | 3 years

SECONDARY OUTCOMES:
To confirm the protection against polio among the Swedish population by measuring antibody levels in serum using NT against Polio virus types 1-3 | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Rigmor Thorstensson, Assoc. Prof., Study Director — Swedish Institute for Infectious Disease Control; Eva Netterlid, Principal Investigator — Swedish Institute for Infectious Disease Control
Locations (1):
- Swedish Institute for Infectious Disease Control, Solna, Sweden

REFERENCES:
- [Derived] Hallander HO, Lepp T, Ljungman M, Netterlid E, Andersson M. Do we need a booster of Hib vaccine after primary vaccination? A study on anti-Hib seroprevalence in Sweden 5 and 15 years after the introduction of universal Hib vaccination related to notifications of invasive disease. APMIS. 2010 Nov;118(11):878-87. doi: 10.1111/j.1600-0463.2010.02674.x. Epub 2010 Sep 2. PMID 20955461